CLINICAL TRIAL: NCT03450239
Title: An fMRI Investigation Into Compulsivity in Those Who Have Recovered From Anorexia Nervosa
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Investigation Into Compulsivity in Anorexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R47959/RE004
Record Dates: First submitted 2018-02-15; First posted 2018-03-01 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Anorexia Nervosa in Remission (Disorder); Compulsive Behavior
Keywords: MRI
MeSH Terms: conditions — Compulsive Behavior

STUDY DESIGN:
Intervention Model Description: All participants undero go an MRI scan, complete some questionnaires and two computer tasks. Participants are in two groups: those who have recovered from anorexia nervosa, and healthy control participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovered from anorexia nervosa (Experimental): Women who have recovered from Anorexia Nervosa for over a year. BMI over 18.5, aged 18-40, scores on Eating Disorder Examination (EDE) within 1 standard deviation of the global mean. All these participants undergo an MRI scan.
  Interventions: Other: MRI
- Healthy controls (Experimental): Healthy control women. BMI over 18.5, aged 18-40, scores on EDE within 1 standard deviation of the global mean. All these participants undergo an MRI scan.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI scan, including structural imaging, functional imaging (both task-related and structural), and Magnetic Resonance Spectroscopy.

SUMMARY:
The investigators will examine compulsivity in those who have recovered from anorexia nervosa, using a multi-modal MRI study. The neural activation of key fronto-striatal areas will be explored using a task which examines set-shifting and reversal-learning, two key components of compulsivity. Additionally, the functional networks displayed during resting-state MRI will be examined between groups, as will the neurochemicals present (using Magnetic Resonance spectroscopy).

DETAILED DESCRIPTION:
The investigators will perform four different MRI (Magnetic Resonance Imaging) scans during one scanning session on those who have recovered from anorexia nervosa (AN) and healthy controls.

Participants will come to the Warneford hospital for a 2.5 hour screening visit, which will consist of questionnaires and interviews to determine their medical and psychiatric history and current mood, along with a practice of the task they'll do in the scanner. Participants will also complete two tasks which measure compulsivity and can be correlated with their brain activity in the scans. The investigators will also go through a scanning safety form with participants at this time.

Participants will also attend a scanning visit, which will last 1.5 hours. One of the scans will look at how the brain responds to a particular task. This task will examine aspects of compulsivity (which is rigidly repeating actions that aren't rewarding) by using face and house stimuli (see reference 1).

The investigators will also perform a scan when participants are at rest, in order to see if there are differences in the way areas of the brain connect to each other who used to have AN. The scientific literature indicates that there may be differences in the some key brain networks, including one which is thought to be involved in reflection and the self (the default mode network), which might also be linked to compulsivity (see reference 2).

This study will also further investigate some initial pilot findings using Magnetic Resonance Spectroscopy, which allows researchers to examine the levels of different neurochemicals in the brain. It has been found that those with a current diagnosis of AN have lower levels of glutamate (a key brain chemical) compared to healthy controls, which is a finding we seek to extend in those who have recovered from AN (see reference 3).

Aims: The investigators aim to see whether there are differences in the brains of those who have recovered from anorexia compared to those who have never had an anorexia diagnosis. This will be both at rest, and whilst participants are doing a task which measures compulsivity, as compulsivity is thought to be a particular risk factor for eating disorders.

Value: If the investigators are able to identify differences, these might reflect underlying risk factors for eating disorders, which could lead to potential future treatments or prevention schemes.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* BMI over 18.5 and has remained so for the last year
* Score lower than mean+1 standard deviation of global mean scores for young women on the EDE
* Fluent English speaker
* Former diagnosis of anorexia nervosa in relevant group

Exclusion Criteria:

* Any current diagnosis of a psychiatric disorder which in the investigator's opinion could impact study results (e.g. significant depression, anxiety or OCD).
* Any current psychotropic medications.
* Eyesight problems that would prohibit participating in a task-fMRI study.
* Current regular cigarette smoking of over 5 cigarettes per day.
* Recent use of illicit drugs.
* Alcohol intake which indicates an element of alcohol abuse; or unwillingness to refrain from drinking the night before the study visit.
* Any contraindications to MRI scanning (including claustrophobia).
* Participant is pregnant or breast-feeding.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen-Level Dependent (BOLD) signal whilst performing set-shifting and reversal-learning | 1 day (During MRI scan)
  BOLD signal differences between groups during the set-shifting and reversal-learning elements of a task: will be examined in orbitofrontal cortex, dorsolateral prefrontal cortex, and striatum. Analyse using a repeated measures ANOVA with region as within-subject factor and group as between-subject factor. Follow up significant interactions with paired t-tests.

SECONDARY OUTCOMES:
Differences between groups in the connectivity of the fronto-parietal and default mode networks using independent components analysis, dual regression and permutation testing across the brain. | 1 day (During MRI scan)
  A resting state scan will be performed, and an Independent Components Analysis will be performed to identify networks. Dual regression using fronto-parietal and default mode network to test whether there are group differences. This procedure regresses the group-spatial-maps into each subject's 4D dataset to give a set of timecourses, then regresses these timecourses into the same 4D dataset to get a subject-specific set of spatial maps. Then, the researchers will compare the spatial maps across groups of subjects to look for group differences in connectivity across the brain, using randomise permutation testing.
The correlation of the default mode network and frontoparietal network activity with perseverative errors on the Wisconsin Card Sorting Task across groups | 1 day (During MRI scan)
  Correlate perseverative errors on Wisconsin Card Sorting Task with connectivity level of Default Mode Network (DMN) and frontoparietal network
Investigate a difference in levels of glutamate between groups | 1 day (During MRI scan)
  Concentration of cortical glutamate in those who have recovered from anorexia relative to controls. Will be analysed using LCModel to quantify metabolites, then an independent samples t-test.
Examine differences between groups on an impulsivity measure | 1 day (During MRI scan)
  Differences between scores on the Affective Go/No-Go Task. Analysed using a independent-samples t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Cowen, Prof, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chamberlain SR, Menzies L, Hampshire A, Suckling J, Fineberg NA, del Campo N, Aitken M, Craig K, Owen AM, Bullmore ET, Robbins TW, Sahakian BJ. Orbitofrontal dysfunction in patients with obsessive-compulsive disorder and their unaffected relatives. Science. 2008 Jul 18;321(5887):421-2. doi: 10.1126/science.1154433. PMID 18635808
- [Background] Boehm I, Geisler D, King JA, Ritschel F, Seidel M, Deza Araujo Y, Petermann J, Lohmeier H, Weiss J, Walter M, Roessner V, Ehrlich S. Increased resting state functional connectivity in the fronto-parietal and default mode network in anorexia nervosa. Front Behav Neurosci. 2014 Oct 2;8:346. doi: 10.3389/fnbeh.2014.00346. eCollection 2014. PMID 25324749
- [Background] Godlewska BR, Pike A, Sharpley AL, Ayton A, Park RJ, Cowen PJ, Emir UE. Brain glutamate in anorexia nervosa: a magnetic resonance spectroscopy case control study at 7 Tesla. Psychopharmacology (Berl). 2017 Feb;234(3):421-426. doi: 10.1007/s00213-016-4477-5. Epub 2016 Dec 1. PMID 27909746